CLINICAL TRIAL: NCT00815997
Title: Novel Angioplasty USIng Coronary Accessor
Acronym: NAUSICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NAUSICA Investigators (Network)
Collaborators: NPO International TRI Network (Network)
Responsible Party: Principal Investigator, Shigeru Saito, Vice President, Shonan Kamakura Genaral Hospital, NAUSICA Investigators
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-28
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Patency of the Radial Artery
Keywords: radial artery; transradial intervention; stent
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6-Fr TRI (transradial coronary intervention) (Sham Comparator): TRI will be performed using a 6-Fr guiding catheter.
  Interventions: Procedure: PCI (percutaneous coronary intervention)
- 4-Fr TRI (Active Comparator): TRI will be performed using a 4-Fr guiding catheter.
  Interventions: Procedure: PCI (percutaneous coronary intervention)

INTERVENTIONS:
Procedure: PCI (percutaneous coronary intervention) — PCI will be performed via the radial artery.

SUMMARY:
To investigate the advantage of using a 4Fr guiding catheter over a 6 Fr, frequencies of radial artery occlusion after transradial coronary intervention (TRI) will be evaluated. Radial artery occlusion rate in 4 Fr TRI group is expected to be not more than that in 6Fr groups.

DETAILED DESCRIPTION:
Prerequisites for TRI were a sufficiently pulsating radial artery and presence of an ulnar pulse with a sufficient palmar arch, as evidenced by the absence of digital ischemia according to the Allen's test. Exclusion criteria for the current study included planned use of a cutting balloon, rotational atherectomy, directional coronary atherectomy, and intravascular ultrasound, which were not compatible with 4-Fr catheter.

Patency of the radial artery after TRI will be evaluated by pulsation of the radial artery, and frequencies of which will be compared between those receiving 4Fr vs 6 Fr coronary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Prerequisites for transradial intervention were a sufficiently pulsating radial artery and presence of an ulnar pulse with a sufficient palmar arch, as evidenced by the absence of digital ischemia according to the Allen's test.

Exclusion Criteria:

* Exclusion criteria included planned use of a cutting balloon, rotational atherectomy, directional coronary atherectomy, and intravascular ultrasound, which were not compatible with 4-Fr catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-01-01; Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Vice Preseident, Shonan Kamakura General Hospital
Locations (19):
- India (2):
  - Global Hospital, Hyderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences, Secunderabad, Andhra Pradesh
- Japan (16):
  - Tosei General Hospital, Seto, Aichi-ken
  - Chibaken Saiseikai Narashino Hospital, Narashino, Chiba
  - Shin-Koga Hospital, Kurume, Fukuoka
  - Kin-ikyo Central Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Sakurakai Takahashi Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Shonan Atsugi Hospital, Atsugi, Kanagawa
  - Tokai University, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kumamoto Rosai Hospital, Yatsushiro, Kumamoto
  - Jichi Medical University, Shimotsuke, Tochigi
  - Aomori Prefectural Central Hospital, Aomori
  - Fukuoka Heart Clinic, Fukuoka
  - Kyoto Kujo Hospital, Kyoto
- Cheng Hsin General Hospital, Taipei, Pai-Tou, Taiwan

REFERENCES:
- [Derived] Takeshita S, Asano H, Hata T, Hibi K, Ikari Y, Kan Y, Katsuki T, Kawasaki T, Masutani M, Matsumura T, Premchand RK, Rao SP, Suzuki T, Takahashi A, Takeda R, Tanaka S, Yamazaki S, Yin WH, Yoshimachi F, Saito S; NAUSICA Trial Investigators. Comparison of frequency of radial artery occlusion after 4Fr versus 6Fr transradial coronary intervention (from the Novel Angioplasty USIng Coronary Accessor Trial). Am J Cardiol. 2014 Jun 15;113(12):1986-9. doi: 10.1016/j.amjcard.2014.03.040. Epub 2014 Apr 1. PMID 24786357

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 Fr TRI: TRI will be performed using a 6-Fr guiding catheter.
Period: Overall Study
Arm/Group | 6 Fr TRI | 4-Fr TRI
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The trial was powered to show the noninferiority of 4-Fr compared with 6-Fr in achieving the primary endpoint of radial artery patency, with a 2-sided alpha level of 0.05. Assuming a radial artery occlusion rate of 1% in the 4-Fr and 6% in the 6-Fr, with a noninferiority margin, δ, of 5%.
Groups:
- 4-Fr TRI: TRI will be performed using a 4-Fr guiding catheter.
  TRI using a 4-Fr guiding catheter: TRI will be performed using a 4-Fr guiding catheter.
- Total: Total of all reporting groups
Arm/Group | 6 Fr TRI | 4-Fr TRI | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 38 | 70
  >=65 years | 48 | 42 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11) | 68 (11) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 18 | 23
  Male | 75 | 62 | 137
Region of Enrollment [Number; unit: participants]
  Taiwan | 12 | 10 | 22
  Japan | 61 | 60 | 121
  India | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Radial Artery Occlusion
Description: The primary endpoint was radial artery occlusion the day after TRI, defined as the absence of a radial pulse confirmed by a reverse Allen's test.
Time Frame: within 2 days after TRI
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Fr TRI | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
Participants | 3 | 0

2. Secondary Outcome: Number of Patients With Successful PCI
Description: Procedural success was defined as a postprocedural residual stenosis of less than 20%, and a thrombolysis in myocardial infarction (TIMI) grade 3 angiographic flow without MACE during in-hospital follow-up.
Time Frame: within 2 days after TRI
Measure: Number; unit: participants
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
participants | 79 | 79

3. Secondary Outcome: Number of Patients With Measure Adverse Cardiac Event (MACE)
Description: Defined as a composite of cardiac death, myocardial infarction, and target lesion revascularization
Time Frame: within 2 days after TRI
Measure: Number; unit: participants
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
participants | 0 | 0

4. Secondary Outcome: Number of Patients With Access-site Complications
Description: Access-site-related complications were defined as bleeding, pseudoaneurysm, arteriovenous fistula, and occlusion of the radial artery, which were considered to be major if they were associated with a vascular repair or a blood transfusion.
Time Frame: within 2 days after TRI
Measure: Count of Participants; unit: Participants
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
Participants | 5 | 0

5. Secondary Outcome: Fluoroscopy Time Used for the Procedure
Description: Fluoroscopy time used for the procedure (minutes).
Time Frame: At the end of TRI
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
minutes | 12 (11) | 13 (9)

6. Secondary Outcome: Contrast Dye Volume Used for the Procedure
Description: Contrast dye volume used for the procedure (mL).
Time Frame: At the end of TRI
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
mL | 101 (68) | 87 (45)

7. Secondary Outcome: Time Used for the Procedure
Description: Time used for the procedure (minutes).
Time Frame: At the end of TRI
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
minutes | 37 (22) | 37 (21)

8. Secondary Outcome: Time Used for Hemostasis
Description: Time Used for Hemostasis (minutes).
Time Frame: within 2 days afterTRI
Measure: Mean (Standard Error); unit: minutes
Arm/Group | 6-Fr TRI (Transradial Coronary Intervention) | 4-Fr TRI
Number analyzed (Participants) | 80 | 80
minutes | 320 (238) | 237 (105)

ADVERSE EVENTS:
Arm/Group | 6 Fr TRI | 4-Fr TRI
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes